CLINICAL TRIAL: NCT04264468
Title: Correlation Between Molecular Typing and Neoadjuvant Chemotherapy in Breast Cancer Patients Based on Mammaprint/Blueprint Test
Acronym: CMTNCMB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMTNCMB
Record Dates: First submitted 2020-01-29; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Evaluation of the Value of Mammaprint Test Gene Variation in the Prediction of Neoadjuvant Chemotherapy for Breast Cancer
Keywords: neoadjuvant chemotherapy; Mammaprint; blueprint; prognosis
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- response group and the non-response group: Received neoadjuvant chemotherapy according to the routine clinical diagnosis and treatment, and evaluated the clinical efficacy once every two cycles of chemotherapy. According to the clinical efficacy, the patients were divided into the neoadjuvant chemotherapy response group and the non-response group (evaluation standard RECIST1.1).
  Interventions: Combination Product: neoadjuvant chemotherapy

INTERVENTIONS:
Combination Product: neoadjuvant chemotherapy — This study prospectively included 150 breast cancer patients (30 patients in the first stage and 120 patients in the second stage) who were treated with the commonly used neoadjuvant chemotherapy recommended by NCCN, received surgical treatment after neoadjuvant chemotherapy, and evaluated the efficacy according to the surgical pathological response.Based on the Mammaprint technology analysis of patients with pathologic complete response (pCR), partial response and no response, we analyzed the characteristic genes related to breast cancer in the tumor tissues and evaluated the accuracy and sensitivity of the Mammaprint test for the efficacy of neoadjuvant chemotherapy

SUMMARY:
This study prospectively included 150 breast cancer patients (30 patients in the first stage and 120 patients in the second stage) who were treated with the commonly used neoadjuvant chemotherapy recommended by NCCN, received surgical treatment after neoadjuvant chemotherapy, and evaluated the efficacy according to the surgical pathological response.Based on the technical analysis of Mammaprint in patients with pathologic complete response (pCR), partial response and no response, we analyzed the characteristic genes related to breast cancer in tumor tissues and evaluated the accuracy and sensitivity of Mammaprint test in the efficacy of neoadjuvant chemotherapy.A new model for predicting NCT effect of breast cancer with combined risk genes and clinical parameters was established based on the clinical characteristic parameters of patients to study the accuracy and sensitivity of Mammaprint monitoring for prognosis determination of breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed new breast cancer (invasive cancer)
* Clinical stage II-III
* women
* Aged 25-80
* At least 6 months of follow-up data, clinical diagnosis and treatment information and personal information available for follow-up are complete
* Complete biological samples required for the study: fresh/frozen tissues/white tablets/wax blocks meeting the requirements of the experiment (before neoadjuvant chemotherapy)
* Tumor markers and imaging data were complete
* Neoadjuvant chemotherapy is commonly recommended by the standard NCCN guidelines

Exclusion Criteria:

* Subjects refuse to participate
* First diagnosis of stage I or IV breast cancer
* Pathological diagnosis of concurrent (or previous) other malignant tumors
* Prehistory breast cancer
* Younger than 25 or older than 80
* Clinical diagnosis and treatment information or biological samples required by the research institute do not meet the needs of the experiment

Ages: 25 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women
Study Population: * Pathologically confirmed new breast cancer (invasive cancer)
  * Clinical stage II-III
  * women
  * Aged 25-80
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-05-14 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence Score variation after neoadjuvant chemotherapy | 6 months
  The recurrence score of each subtype

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China